CLINICAL TRIAL: NCT01885481
Title: Evaluation of Efficacy and Safety of Epidural Steroid Injection Using Dexamethasone or Betamethasone in Patients With Spinal Pain: a Prospective, Randomized, Double-blind Study
Brief Title: Evaluation of Efficacy and Safety of Epidural Steroid Injection Using Dexamethasone or Betamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Joon Woo Lee, Associate professor, Department of Radiology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1304-199-001
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Back Pain; Neck Pain
Keywords: dexamethasone; betamethasone; epidural steroid injection; comparative effectiveness research
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Dexamethasone; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESI-1 (Active Comparator): epidural steroid injection using dexamethasone
  Interventions: Drug: Dexamethasone
- ESI-2 (Experimental): epidural steroid injection using betamethasone
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Dexamethasone — epidural steroid injection using dexamethasone
  Other Names: dexamethasone-ESI
  Arms: ESI-1
Drug: Betamethasone — epidural steroid injection using betamethasone
  Other Names: betamethasone-ESI
  Arms: ESI-2

SUMMARY:
Particle steroid drug such as triamcinolone has been used widely for epidural steroid injection (ESI) treatment in Korea. However, Korea FDA recently prohibit ESI using triamcinolone, following the regulation of US FDA. Therefore, dexamethasone and betamethasone become only candidate drugs for ESI in Korea and the investigators are curious about the effectiveness and safety of both drugs due to limitation of information about comparison of two drugs in previous literature. So, this study aims to compare the effectiveness and safety of both drugs and our hypothesis is that there is no difference of the effectiveness between dexamethasone and betamethasone at 2 weeks after ESI.

ELIGIBILITY:
Inclusion Criteria:

1. patients with spinal pain (i.e.neck pain, back pain, or radiculopathy..)
2. patients with informed consent
3. visual analog scale (VAS) is five or more in 10-point scale at screening
4. sustained spinal pain, regardless of sufficient conservative treatment (i.e. oral medicine, physical therapy..)

Exclusion Criteria:

1. age of patient less than 19 years
2. relative contraindication of epidural steroid injection, as follows:

   * pregnant or breast-feeding state
   * uncontrolled coagulopathy
   * suspected of active infection state
   * uncontrolled diabetes mellitus
   * previous history of adverse event related to epidural steroid injection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with pain improvement | baseline and 2 weeks
  the proportion of patients with significant pain improvement at 2 week after epidural steroid injection, with the patients' subjective satisfaction scale of "much improved" or "no pain"

SECONDARY OUTCOMES:
incidence of adverse events | during 12 weeks after epidural steroid injection
  incidence of adverse event during 12 weeks after epidural steroid injection
pain relief | baseline and 2 weeks
  decrease of visual analog scale (VAS) for pain at 2 week time point after epidural steroid injection, compared to baseline at 0 week
disability improvement | baseline and 2 weeks
  decrease of disability index (Oswestry disability index or Neck disability index) for pain at 2 week time point after epidural steroid injection, compared to baseline at 0 week

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Lee, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No